CLINICAL TRIAL: NCT06702449
Title: A Seamless Phase 1/2, Observer-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Safety and Immunogenicity of a UTI Vaccine When Administered to Adults 18 Through 64 Years of Age and Clinical Efficacy When Administered to Females 18 Through 64 Years of Age
Brief Title: A Study on the Safety and Immune Response of a Urinary Tract Infection (UTI) Vaccine in Adults 18-64 Years of Age and Clinical Efficacy in Females 18-64 Years of Age
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 219685
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Tract infection (UTI); UTI vaccine; E. coli; Safety; Immunogenicity; Efficacy
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1 Group A1/A2 (Experimental): Participants receive candidate UTI vaccine low dose formulation 1 or placebo on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine low dose formulation 1; Combination Product: Placebo
- Part 1 Group B1/B2 (Experimental): Participants receive candidate UTI vaccine low dose formulation 2, or placebo on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine low dose formulation 2; Combination Product: Placebo
- Part 1 Group C1/C2 (Experimental): Participants receive candidate UTI vaccine medium dose formulation 1, or placebo on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine medium dose formulation 1; Combination Product: Placebo
- Part 1 Group D1/D2 (Experimental): Participants receive candidate UTI vaccine medium dose formulation 2, or placebo on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine medium dose formulation 2; Combination Product: Placebo
- Part 1 Group E1/E2 (Experimental): Participants receive candidate UTI vaccine high dose formulation 1, or placebo on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine high dose formulation 1; Combination Product: Placebo
- Part 1 Group F1/F2 (Experimental): Participants receive candidate UTI vaccine high dose formulation 2, or placebo on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine high dose formulation 2; Combination Product: Placebo
- Part 2 Group 1 (Experimental): Participants receive the candidate UTI vaccine highest tolerated dose (HTD) formulation 2, tested in Part 1 of the study, on Day 1 and Day 61.
  Interventions: Combination Product: Candidate UTI vaccine HTD formulation 2
- Part 2 Group 2 (Placebo Comparator): Participants receive placebo on Day 1 and Day 61.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Candidate UTI vaccine low dose formulation 1 — Candidate UTI vaccine low dose formulation 1 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group A1/A2
Combination Product: Candidate UTI vaccine low dose formulation 2 — Candidate UTI vaccine low dose formulation 2 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group B1/B2
Combination Product: Candidate UTI vaccine medium dose formulation 1 — Candidate UTI vaccine medium dose formulation 1 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group C1/C2
Combination Product: Candidate UTI vaccine medium dose formulation 2 — Candidate UTI vaccine medium dose formulation 2 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group D1/D2
Combination Product: Candidate UTI vaccine high dose formulation 1 — Candidate UTI vaccine high dose formulation 1 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group E1/E2
Combination Product: Candidate UTI vaccine high dose formulation 2 — Candidate UTI vaccine high dose formulation 2 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group F1/F2
Combination Product: Candidate UTI vaccine HTD formulation 2 — Candidate UTI vaccine HTD formulation 2 administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 2 Group 1
Combination Product: Placebo — Placebo administered intramuscularly according to a 0, 2 months administration schedule.
  Arms: Part 1 Group A1/A2; Part 1 Group B1/B2; Part 1 Group C1/C2; Part 1 Group D1/D2; Part 1 Group E1/E2; Part 1 Group F1/F2; Part 2 Group 2

SUMMARY:
The purpose of this study is to assess safety, reactogenicity, and immune response of the candidate UTI vaccine compared to placebo in adults between and including 18-64 years of age (YOA), and to perform a preliminary evaluation of clinical efficacy in females between and including 18-64 YOA.

DETAILED DESCRIPTION:
This clinical trial consists of 2 parts. Part 1 will consist of antigen dose-escalation (start with least dose with gradual increase in dose) Safety Lead-In (SLI) in healthy participants. Part 2 (Proof of Principle [PoP]) will start after the safety review of all safety data in Part 1 and will consist of participants with history of at least 1 episode of urine culture confirmed E. coli UTI in the last 12 months prior to the study intervention administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Female participants of non-childbearing potential may be enrolled in the clinical study.
* Female participants of childbearing potential may be enrolled in the clinical study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for at least 1 month after completion of the study intervention administration series.
* Blood sample for simultaneous follicle stimulating hormone (FSH) and estradiol levels may be collected.

Additional inclusion criterion only for participants in Part 1 of the study (SLI):

* Female and male between and including 18 through 64 YOA at the time of ICF signature.
* Healthy participants, according to medical history, laboratory assessment and clinical examination at Screening Visit.

Additional inclusion criterion only for participants in Part 2 of the study (PoP):

* Females between and including 18 through 64 YOA at the time of ICF signature.
* Female participants with documented history of at least 1 episode of urine culture confirmed E. coli uncomplicated UTI in the last 12 months prior to study vaccine administration.

Exclusion Criteria:

Medical conditions:

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity to latex.
* History of pIMD.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* History of endocrinologic, hematologic, metabolic, urologic, dermatologic, or gastrointestinal conditions that, in the opinion of the investigator, places the participant at unacceptable risk or would make adhering to study procedures for the duration of the study difficult.
* Recurrent history or uncontrolled neurological disorders or any neuroinflammatory (including, but not limited to demyelinating disorders, encephalitis or myelitis of any origin), congenital neurological conditions, encephalopathies, or seizures.
* Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study.
* Condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Additional exclusionary medical conditions only for participants in Part 1 of the study (SLI):

• Any clinically significant hematologic and/or biochemical laboratory abnormality at Screening Visit.

Additional exclusionary medical conditions only for participants in Part 2 of the study (PoP):

* The participant has UTI that is known or suspected to be due to fungal, parasitic, or viral pathogens; or known or suspected to be due to Pseudomonas aeruginosa or any Enterobacter species.
* The participant has symptoms known or suspected to be caused by another disease process, such as asymptomatic bacteriuria, overactive bladder, chronic incontinence, or chronic interstitial cystitis, that may interfere with the clinical efficacy assessments.
* The participant has an anatomical or physiological anomaly that predisposes the participant to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction or stricture of the urinary tract, primary renal disease or neurogenic bladder, or the participant has a history of anatomical or functional abnormalities of the urinary tract.
* The participant has an indwelling catheter, nephrostomy, ureteral stent, or other foreign material in the urinary tract.
* The participant who, in the opinion of the investigator, has an otherwise complicated UTI or has an active upper UTI.
* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention(s) during the period beginning 30 days before the first dose of study intervention(s) (Day -29 to Day 1), or their planned use during the study period.
* Previous administration of a vaccine or immunostimulant targeting rUTI.
* Participants currently on a prophylactic agent for rUTI (including antibiotics, methenamine, D-mannose).
* Planned administration and/or administration of a vaccine not foreseen by the study protocol in the period starting 15 days before the first dose and ending 15 days after the last dose of study intervention(s) administration.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the study intervention or planned administration during the study period.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune modifying treatments at any time up to the end of the study.

  * Up to 3 months prior to the study intervention administration:
  * For corticosteroids, this will mean prednisone equivalent >=20 mg/day for adult participants. Inhaled and topical steroids are allowed.
  * Up to 3 months prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug, vaccine or invasive medical device).
* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions before 1 month after completion of the study intervention administration series.
* History of chronic alcohol consumption and/or drug abuse, based on investigator judgment.
* Persons under guardianship or trusteeship.
* Persons deprived of liberty.
* Any study personnel or their immediate dependents, family, or household members.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 448 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Number of participants reporting solicited administration site adverse events (AEs) | During the 7 days follow-up period post-Dose 1 (study intervention administered at Day 1)
  Solicited administration site events include pain, redness and swelling at administration site.
Part 1 and 2: Number of participants reporting solicited administration site AEs | During the 7 days follow-up period post-Dose 2 (study intervention administered at Day 61)
  Solicited administration site events include pain, redness and swelling at administration site.
Part 1 and 2: Number of participants reporting solicited systemic AEs | During the 7 days follow-up period post-Dose 1 (study intervention administered at Day 1)
  Solicited systemic events include fever, headache, myalgia (muscle pain), arthralgia (joint pain), and fatigue (tiredness). Fever is defined as temperature greater than or equal to (>=) 38.0°C and preferred location for measuring temperature is the axilla.
Part 1 and 2: Number of participants reporting solicited systemic AEs | During the 7 days follow-up period post-Dose 2 (study intervention administered at Day 61)
  Solicited systemic events include fever, headache, myalgia (muscle pain), arthralgia (joint pain), and fatigue (tiredness). Fever is defined as temperature >=38.0°C and preferred location for measuring temperature is the axilla.
Part 1 and 2: Number of participants reporting unsolicited AEs | During the 30 days follow-up period post-Dose 1 (study intervention administered at Day 1)
  An unsolicited AE is an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Part 1 and 2: Number of participants reporting unsolicited AEs | During the 30 days follow-up period post-Dose 2 (study intervention administered at Day 61)
  An unsolicited AE is an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Part 1 and 2: Number of participants reporting any immediate unsolicited AEs | During the 60 minutes follow-up period post-Dose 1 (study intervention administered at Day 1)
  An unsolicited AE is an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Part 1 and 2: Number of participants reporting any immediate unsolicited AEs | During the 60 minutes follow-up period post-Dose 2 (study intervention administered at Day 61)
  An unsolicited AE is an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Part 1 and 2: Number of participants reporting serious adverse events (SAEs) | From Day 1 (Dose 1 administration) until Day 426 (end of follow-up)
  An SAE is defined as any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongs existing hospitalization, results in disability/incapacity or other medically significant events.
Part 1 and 2: Number of participants reporting potential immune-mediated diseases (pIMDs) leading to study withdrawal | From Day 1 (Dose 1 administration) until Day 426 (end of follow-up)
  pIMDs are a subset of Adverse Events of Special Interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Part 1 and 2: Number of participants reporting medically-attended adverse events (MAAEs) leading to study withdrawal | From Day 1 (Dose 1 administration) until Day 426 (end of follow-up)
  An MAAE is defined as an unsolicited AE, such as a symptom or illness, which required hospitalization, or emergency room visit, or visit to/by a health care provider.
Part 1 and 2: Number of participants reporting AEs leading to study withdrawal | From Day 1 (Dose 1 administration) until Day 426 (end of follow-up)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Part 1: Number of participants with hematology or biochemistry abnormalities or changes in baseline value | At 7 days post-Dose 1 (Day 8) compared with baseline (pre-Dose 1, Day 1)
Part 1: Number of participants with hematology or biochemistry abnormalities or changes in baseline value | At 7 days post-Dose 2 (Day 68) compared with Day 61 (pre-Dose 2)
Part 2: Incidence rate (IR) of the first occurrence of a urine culture confirmed UTI due to E. coli in the investigational group compared to the IR in placebo group | From 14 days (Day 75) up to 12 months (Day 426) post-Dose 2

SECONDARY OUTCOMES:
Part 2: IR of the total number of occurrences of urine culture confirmed UTIs due to E. coli in the investigational group compared to the IR in placebo group | From 14 days (Day 75) up to 12 months (Day 426) post-Dose 2
Part 2: IR of the first occurrence of a urine culture confirmed UTI due to E. coli in the investigational group compared to the IR in placebo group | From 14 days post-Dose 1 (Day 15) and up to the day before administration of Dose 2 (Day 60) or, for participants receiving only Dose 1, up to the end of the study (Day 426)
Part 2: IR of the total number of occurrences of urine culture confirmed UTIs due to E. coli in the investigational group compared to the IR in placebo group | From 14 days post-Dose 1 (Day 15) and up to the day before administration of Dose 2 (Day 60) or, for participants receiving only Dose 1, up to the end of the study (Day 426)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Secaucus, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Weatherford, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Wenatchee, Washington
- South Africa (2):
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Soshanguve

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf